CLINICAL TRIAL: NCT01592071
Title: Eliminating IgG-mediated Reactive Foods From the Diet and Its Effect on Body Composition and Quality of Life in Overweight Persons
Brief Title: IgG-mediated Food Test for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Immuno Laboratories (Unknown)
Responsible Party: Principal Investigator, John E. Lewis, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20080670
Record Dates: First submitted 2012-05-01; First posted 2012-05-07 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Overweight and Obesity
Keywords: food sensitivity; IgG; obesity; overweight; body composition; reactive foods
MeSH Terms: conditions — Overweight; Obesity; Food Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Replace reactive w/ non-reactive foods (Experimental): Test results, individual dietary plan: 'Replace reactive foods with non-reactive foods'
  Interventions: Other: Replace reactive foods with non-reactive foods

INTERVENTIONS:
Other: Replace reactive foods with non-reactive foods — Subjects were provided with the test results and an individualized dietary plan based on replacing reactive foods with non-reactive foods as replacements per the Immuno Bloodprint results.

SUMMARY:
This study assessed the effect of an IgG-mediated food sensitivity test in combination with a food elimination diet on body composition and secondary outcomes in people who were overweight.

DETAILED DESCRIPTION:
This study looked at foods that stimulated IgG food antibody production, which may play a role in certain conditions, such as irritable bowel syndrome, obesity, type I diabetes, and migraine headaches.

Using a proprietary blood test, the Immuno Bloodprint, to determine which foods stimulate IgG food antibodies in each person, this study detailed a personalized list of reactive foods that stimulated such antibodies for each participant. The participant was then advised to eliminate as much as possible the reactive foods for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI above 20
* Express an interest in losing weight

Exclusion Criteria:

* Less than 18 years of age
* Currently participating in another research trial for weight loss
* Suffering from serious medical complications that might limit their participation, such as recent heart attack, stroke, or chronic kidney disease
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Lewis, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami CRB, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between 2008 and 2010. Blood draws and discussion of results of blood draws performed at UM Clinical Research Building
Groups:
- Non-reactive Foods: Subjects had blood drawn for proprietary test known as the Immuno Bloodprint. Subjects were provided with the test results and an individualized dietary plan based on replacing reactive foods with non-reactive foods as replacements. The primary advice to each participant was to focus as much as possible on eliminating the reactive foods from the diet for a 90-day period.
Period: Overall Study
Arm/Group | Non-reactive Foods
Started | 120
Completed | 120
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 116
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Weight (kg)
Description: Measure of body composition: weight (kg).
Time Frame: 30, 60 and 90 days from baseline
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
kilograms
  Weight (Baseline) | 80 (17.2) [2.1 to 5.2]
  Weight (30 days) | 76.6 (15.8) [2.6 to 7.5]
  Weight (60 days) | 74.7 (16) [1.7 to 9.4]
  Weight (90 days) | 75 (17.7)

2. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure measured.
Time Frame: 30, 60 and 90 days from baseline
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
mm Hg
  Systolic BP (Baseline) | 123.2 (17.2)
  Systolic BP (30 days) | 119.0 (12.7)
  Systolic BP (60 days) | 119.0 (15.1)
  Systolic BP (90 days) | 115.7 (13.7)
  Diastolic BP (Baseline) | 79.0 (12.1)
  Diastolic BP (30 days) | 75.9 (9.1)
  Diastolic BP (60 days) | 75.0 (9.6)
  Diastolic BP (90 days) | 74.0 (7.3)

3. Primary Outcome: Body Mass Index
Description: Measure of body composition: height and weight to assess BMI.
Time Frame: 30, 60 and 90 days from baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
kg/m^2
  BMI (Baseline) | 29.0 (5.5) [0.38 to 0.93]
  BMI (30 days) | 27.7 (5.6) [0.57 to 1.37]
  BMI (60 days) | 27.4 (5.6) [0.46 to 1.67]
  BMI (90 days) | 27.2 (5.6)

4. Primary Outcome: Waist Circumference
Description: Measure of body composition: waist circumference (cm).
Time Frame: 30, 60 and 90 days from baseline
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
centimeters
  Waist Circumference (Baseline) | 91.7 (14.5)
  Waist Circumference (30 days) | 85.9 (12.7)
  Waist Circumference (60 days) | 85.1 (11.7)
  Waist Circumference (90 days) | 84.3 (12.4)

5. Secondary Outcome: Heart Rate
Description: Heart rate measured.
Time Frame: 30, 60 and 90 days from baseline
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
bpm
  Heart Rate (Baseline) | 73.6 (10.7)
  Heart Rate (30 days) | 72.1 (9.9)
  Heart Rate (60 days) | 73.3 (8.9)
  Heart Rate (90 days) | 72.5 (8.4)

6. Secondary Outcome: Quality of Life
Description: Quality of life categories measured with the SF-36 Health Survey. The SF-36 Health Survey provides psychometrically-based physical and mental health summary measures and a preference-based health utility index.The SF-36 provides a t-score for each scale or domain ranging from 0-100 with higher scores representing better perceived quality of life.
Time Frame: 30, 60 or 90 days from baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
Scores on a scale
  Physical Functioning (Baseline) | 86.5 (17.9) [-10.8 to -0.23]
  Physical Functioning (30 days) | 91.8 (11.5) [-13.0 to -3.8]
  Physical Functioning (60 days) | 91.7 (9.9) [-17.1 to -5.9]
  Physical Functioning (90 days) | 93.8 (7.0) [-14.3 to -2.8]
  Physical Role Functioning (Baseline) | 83.9 (21.4) [-14.6 to -1.0]
  Physical Role Functioning (30 days) | 91.6 (16.5) [-12.7 to -3.6]
  Physical Role Functioning (60 days) | 88.3 (14.1) [-20.9 to -6.2]
  Physical Role Functioning (90 days) | 95.6 (6.1) [-18.1 to -2.5]
  Emotional Role Functioning (Baseline) | 85.9 (19.2) [-16.2 to -1.2]
  Emotional Role Functioning (30 days) | 91.7 (16.2) [-22.3 to -5.5]
  Emotional Role Functioning (60 days) | 95.5 (9.5) [-18.3 to -3.4]
  Emotional Role Functioning (90 days) | 93.3 (9.6) [-19.2 to -4.7]
  Mental Health (Baseline) | 75.6 (15.9) [-22.0 to -5.4]
  Mental Health (30 days) | 83.0 (15.1) [-14.0 to -3.9]
  Mental Health (60 days) | 81.7 (12.7) [-15.7 to -2.5]
  Mental Health (90 days) | 86.5 (10.1)
  Social Functioning (Baseline) | 80.1 (22.8)
  Social Functioning (30 days) | 87.5 (20.3)
  Social Functioning (60 days) | 88.5 (14.2)
  Social Functioning (90 days) | 94.4 (10.3)
  Vitality (Baseline) | 57.7 (17.8)
  Vitality (30 days) | 69.9 (16.2)
  Vitality (60 days) | 68.0 (13.7)
  Vitality (90 days) | 70.3 (14.7)
  Bodily Pain (Baseline) | 67.3 (22.3)
  Bodily Pain (30 days) | 78.4 (14.3)
  Bodily Pain (60 days) | 79.4 (9.6)
  Bodily Pain (90 days) | 78.5 (13.6)
  General Health (Baseline) | 70.9 (19.6)
  General Health (30 days) | 82.4 (13.8)
  General Health (60 days) | 79.3 (13.4)
  General Health (90 days) | 81.1 (11.0)

7. Primary Outcome: Hip Circumference
Description: Measure of body composition: hip circumference (cm).
Time Frame: 30, 60 or 90 days from baseline
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
centimeters
  Hip Circumference (Baseline) | 106.4 (11.4)
  Hip Circumference (30 days) | 103.1 (12.4)
  Hip Circumference (60 days) | 103.4 (13.5)
  Hip Circumference (90 days) | 102.9 (11.2)

8. Primary Outcome: Waist-Hip Ratio (WHR)
Description: Measure of body composition: hip and waist circumference to calculate waist/hip ratio (WHR).
Time Frame: 30, 60 or 90 days from baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Non-reactive Foods
Number analyzed (Participants) | 120
ratio
  Waist-Hip Ratio (Baseline) | 0.86 (0.11) [0.1 to 2.57]
  Waist-Hip Ratio (30 days) | 0.84 (0.12) [0.78 to 3.36]
  Waist-Hip Ratio (60 days) | 0.83 (0.09) [0.56 to 3.15]
  Waist-Hip Ratio (90 days) | 0.82 (0.08) [1.38 to 3.33]

ADVERSE EVENTS:
Description: Serious or Other (non-serious) Adverse Events were collected/assessed, but none observed.
Arm/Group | Non-reactive Foods
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No